CLINICAL TRIAL: NCT03185312
Title: Cutaneous JAK Expression in Vitiligo and Acne Vulgaris.
Brief Title: Cutaneous JAK in Vitiligo and Acne Vulgaris.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmin Mostafa Tawfik, lecturer, Assiut University
Other Study IDs: CJEIVAA
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Vitiligo and Acne Vulgaris
MeSH Terms: conditions — Vitiligo; Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with acne vulgaris: Clinical evaluation including full history taking and dermatological examination will be done for all patients. Assessment of disease severity will be performed using Global acne severity grading for acne vulgaris Skin biopsies will be taken from lesional and non-lesional skin .immunohistochemical staining using specific antibodies for detection of expression of JAK1, JAK2 and JAK3.
  Interventions: Diagnostic Test: skin biopsy
- patients with vitiligo: Clinical evaluation including full history taking and dermatological examination will be done . Assessment of disease severity will be performed using VASI score Skin biopsies will be taken from lesional and non-lesional skin .immunohistochemical staining using specific antibodies for detection of expression of JAK1, JAK2 and JAK3..
  Interventions: Diagnostic Test: skin biopsy
- control: Skin biopsies will be taken from skin of controls.
  . Five micron thick sections will be cut from paraffin blocks for immunohistochemical staining using specific antibodies for detection of expression of JAK1, JAK2 and JAK3.
  Interventions: Diagnostic Test: skin biopsy

INTERVENTIONS:
Diagnostic Test: skin biopsy — Clinical evaluation including full history taking and dermatological examination will be done for all patients. Assessment of disease severity will be performed using VASI score for vitiligo and Global acne severity grading for acne vulgaris Skin biopsies will be taken from lesional and non-lesional skin of patients as well as controls. immunohistochemical staining using specific antibodies for detection of expression of JAK1, JAK2 and JAK3.
  Additionally, biopsies will be preserved in RNA later solution at -20°C. RNA isolation and real-time qPCR analysis will be performed for measurement of cutaneous JAK1, JAK2 and JAK3 gene expression.

SUMMARY:
The Janus kinase/signal transducer and activator of transcription (JAK-STAT) cytokine signaling pathway is an emerging area of interest in dermatology, and emerging evidence suggests that this pathway may play a crucial role in pathogenesis of inflammatory skin disorders.

Recent advances on the role of cytokines in the pathophysiology of immune mediated inflammatory diseases lead to the understanding that many pro inflammatory interleukins use JAK/STAT components for signal transduction .

DETAILED DESCRIPTION:
The JAK/STAT signaling pathway transmits information from extracellular chemical signals to the nucleus resulting in DNA transcription. Binding of ligands, such as interferon and interleukins, to their specific transmembrane receptors activate associated JAKs. Phosphorylation of STAT follows, and the phosphorylated STAT translocates to the cell nucleus and activates transcription or suppression of target genes .

The JAK family of non-receptor intracellular tyrosine kinases is comprised of four members, JAK1, JAK2, JAK3 and tyrosine kinase (TyK)2. The JAKs are selectively activated by different receptors and have, therefore, distinct in vivo roles. JAK1 is mainly activated by type II cytokine receptors. JAK2 is crucial in transducing signals for cytokine receptors involved in hematopoiesis (erythropoietin, thrombopoietin and haematopoietic cell development cytokines). JAK3 is mainly expressed in B and T lymphocytes, and TYK2 associates commonly with other JAKs.

Cutaneous JAK overexpression has already been demonstrated in a number of inflammatory skin diseases (ISDs) including psoriasis, lichen planus (LP), atopic dermatitis (AD), pyoderma gangrenosum (PG) and alopecia areata (AA); indicating its crucial role in inflammatory keratinocytes.

Furthermore, the recent discovery of the JAK/STAT signaling pathway opened a new window of opportunity for the treatment of ISDs and promoted the development of drugs that block JAK activation.

JAK inhibitors in oral and topical formulations have shown beneficial results in psoriasis and alopecia areata. Patients suffering from vitiligo might also benefit from JAK inhibition. Recently, significant repigmentation was reported in a patient with vitiligo after treatment with tofacitinib, an oral JAK 1/3 inhibitor . However, the knowledge of the cutaneous JAK involvement in vitiligo is scarce. Similarly, little is known about cutaneous JAK expression in acne vulgaris.

Considering the previous findings, there is a need for further elucidation of the JAK signaling in other skin diseases as vitiligo and acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* patients with vitiligo and acne vulgaris.

Exclusion Criteria:

* patients below 12 years of age, or receiving systemic treatments in the last month

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A group of 20 patients with vitiligo and 20 patients with acne vulgaris and another control group of 20 age and sex matched healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
To analyze the cutaneous JAK expression in vitiligo and acne vulgaris, assess cutaneous JAK expression in relation to disease severity in vitiligo and acne vulgaris compared to controls | 1 year
  Skin biopsies will be taken from lesional and non-lesional skin of patients as well as from healthy volunteers as controls.
  All biopsies will be derived from untreated skin lesions for a minimum of 15 days before the biopsy The biopsies will be fixed and paraffin embedded. Five micron thick sections will be cut from paraffin blocks for immunohistochemical staining using specific antibodies for detection of expression of JAK1, JAK2 and JAK3.
  Additionally, biopsies will be preserved in RNA later solution at -20°C. RNA isolation and real-time qPCR analysis will be performed for measurement of cutaneous JAK1, JAK2 and JAK3 gene expression.

CONTACTS AND LOCATIONS:
Overall Officials: Amira Abdel Motaleb, MD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palanivel JA, Macbeth AE, Chetty NC, Levell NJ. An insight into JAK-STAT signalling in dermatology. Clin Exp Dermatol. 2014 Jun;39(4):513-8. doi: 10.1111/ced.12273. PMID 24825142
- [Background] O'Shea JJ, Murray PJ. Cytokine signaling modules in inflammatory responses. Immunity. 2008 Apr;28(4):477-87. doi: 10.1016/j.immuni.2008.03.002. PMID 18400190
- [Background] Alves de Medeiros AK, Speeckaert R, Desmet E, Van Gele M, De Schepper S, Lambert J. JAK3 as an Emerging Target for Topical Treatment of Inflammatory Skin Diseases. PLoS One. 2016 Oct 6;11(10):e0164080. doi: 10.1371/journal.pone.0164080. eCollection 2016. PMID 27711196
- [Background] Rawlings JS, Rosler KM, Harrison DA. The JAK/STAT signaling pathway. J Cell Sci. 2004 Mar 15;117(Pt 8):1281-3. doi: 10.1242/jcs.00963. No abstract available. PMID 15020666
- [Background] O'Shea JJ, Schwartz DM, Villarino AV, Gadina M, McInnes IB, Laurence A. The JAK-STAT pathway: impact on human disease and therapeutic intervention. Annu Rev Med. 2015;66:311-28. doi: 10.1146/annurev-med-051113-024537. PMID 25587654
- [Background] Damsky W, King BA. JAK inhibitors in dermatology: The promise of a new drug class. J Am Acad Dermatol. 2017 Apr;76(4):736-744. doi: 10.1016/j.jaad.2016.12.005. Epub 2017 Jan 28. PMID 28139263
- [Background] Papp KA, Menter A, Strober B, Langley RG, Buonanno M, Wolk R, Gupta P, Krishnaswami S, Tan H, Harness JA. Efficacy and safety of tofacitinib, an oral Janus kinase inhibitor, in the treatment of psoriasis: a Phase 2b randomized placebo-controlled dose-ranging study. Br J Dermatol. 2012 Sep;167(3):668-77. doi: 10.1111/j.1365-2133.2012.11168.x. PMID 22924949
- [Background] Ports WC, Khan S, Lan S, Lamba M, Bolduc C, Bissonnette R, Papp K. A randomized phase 2a efficacy and safety trial of the topical Janus kinase inhibitor tofacitinib in the treatment of chronic plaque psoriasis. Br J Dermatol. 2013 Jul;169(1):137-45. doi: 10.1111/bjd.12266. PMID 23387374
- [Background] Craiglow BG, King BA. Tofacitinib Citrate for the Treatment of Vitiligo: A Pathogenesis-Directed Therapy. JAMA Dermatol. 2015 Oct;151(10):1110-2. doi: 10.1001/jamadermatol.2015.1520. PMID 26107994
- [Background] Choi JJ, Park MY, Lee HJ, Yoon DY, Lim Y, Hyun JW, Zouboulis CC, Jin M. TNF-alpha increases lipogenesis via JNK and PI3K/Akt pathways in SZ95 human sebocytes. J Dermatol Sci. 2012 Mar;65(3):179-88. doi: 10.1016/j.jdermsci.2011.11.005. Epub 2011 Nov 20. PMID 22305016
- [Derived] Abdel Motaleb AA, Tawfik YM, El-Mokhtar MA, Elkady S, El-Gazzar AF, ElSayed SK, Awad SM. Cutaneous JAK Expression in Vitiligo. J Cutan Med Surg. 2021 Mar-Apr;25(2):157-162. doi: 10.1177/1203475420972340. Epub 2020 Nov 11. PMID 33174479